CLINICAL TRIAL: NCT07135349
Title: A Multi-center, Randomized, Open-label, Phase II Study to Evaluate the Efficacy and Safety of BW-20507 Injection Combined With Pegylated Interferon Alfa in Patients With Chronic Hepatitis B Infection
Brief Title: A Phase II Clinical Study of BW-20507 in Combination With PEG-IFNα for the Treatment of Hepatitis B
Acronym: HBV
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Argo Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BW-20507-2002
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): BW-20507 with/without NUC
  Interventions: Drug: BW-20507 with/without NUC
- Cohort 2 (Experimental): BW-20507 with/without NUC, Peg-IFNa
  Interventions: Drug: BW-20507 with/without NUC, Peg-IFNa

INTERVENTIONS:
Drug: BW-20507 with/without NUC — • BW-20507 with/without NUCs will be administrated for 48 weeks
  Arms: Cohort 1
Drug: BW-20507 with/without NUC, Peg-IFNa — • BW-20507 with/without NUC will be administrated for 48 weeks, Peg-IFNa will be administrated.
  Arms: Cohort 2

SUMMARY:
This is a randomized, open-label, multicenter phase II study to evaluate the efficacy and safety of BW-20507 in combination with PEG-IFNα in CHB patients

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign ICF and are able to complete the procedures as planned for this study.
* Males or females aged 18 to 65 (inclusive) when signing informed consent
* Body mass index (BMI) arranges 18.5 to 32.0 kg/m2 (inclusive)
* Participants must be diagnosed with chronic hepatitis B infection: HBsAg positivity at least 6 months (need documents)
* NUC treatment history and screening status of HBV DNA, HBeAg, HBsAg, and ALT must meet the requirements for different cohorts.
* Males of reproductive potential or females of childbearing potential must agree to utilize reliable contraception, refrain from childbearing plan, and will not donate sperm or eggs during the study

Exclusion Criteria:

* Clinically significant abnormalities
* Significant liver fibrosis or cirrhosis at screening, or a liver stiffness value (LSM) > 9.0 kPa
* Concomitant clinically significant other liver diseases
* Previous/current manifestations of hepatic decompensation
* History of acute or chronic renal insufficiency
* Significant abnormal ECG at screening
* Participants with a history of malignancy or who are being evaluated for a possible malignancy
* Serious mental illness or history
* Thyroid dysfunction or DM
* Suspected history of allergy to any component of the study drug
* Those who are participating in another clinical study, or have not undergone a protocol-specified washout period prior to this study
* Protocol-specified prohibited therapies usage
* Received any antisense oligonucleotides (ASO) or small molecule interfering ribonucleic acid (siRNA) drug
* Any other circumstance or condition that, in the opinion of the investigator, the participants are inappropriate for participation in the study

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-06-07 (Estimated); Study Completion 2028-05-08 (Estimated)

PRIMARY OUTCOMES:
1. The proportion of participants who meet the NUC discontinuation criteria at Week 72 in participants with baseline HBsAg ⩽ 3000 IU/mL and HBeAg-negative. | Week 72

SECONDARY OUTCOMES:
HBsAg changes throughout the study | up to 124 weeks

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Argo Investigative Site, Hefei, Anhui
  - Argo Investigative Site, Beijing, Beijing Municipality
  - Argo Investigative Site, Sichuan, Chengdu
  - Argo Investigative Site, Chongqing, Chongqing Municipality
  - Argo Investigative Site, Fuzhou, Fujian
  - Argo Investigative Site, Guangzhou, Guangdong
  - Argo Investigative Site, Shenzhen, Guangdong
  - Argo Investigative Site, Zunyi, Guizhou
  - Argo Investigative Site, Changzhou, Jiangsu
  - Argo Investigative Site, Xuzhou, Jiangsu
  - Argo Investigative Site, Nanchang, Jiangxi
  - Argo Investigative Site, Jiangxi, Nanchang
  - Argo Investigative Site, Shanghai, Shanghai Municipality
  - Argo Investigative Site, Chengdu, Sichaun
  - Argo Investigative Site, Chengdu, Sichuan
  - Argo Investigative Site, Zhejiang, Wenzhou
  - Argo Investigative Site, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No